CLINICAL TRIAL: NCT01141491
Title: A Randomized, Multicenter, Double-Blind, Phase II Trial of a KLH Conjugated Trivalent Ganglioside Vaccine Containing GM2, GD2 Lactone, and GD3 Lactone With the Immunological Adjuvant OPT-821 Versus OPT-821 Alone in Metastatic Sarcoma Patients Who Are Rendered Disease Free
Brief Title: Trivalent Ganglioside Vaccine With Immunological Adjuvant or Immunological Adjuvant Alone in Metastatic Sarcoma Patients Who Are Rendered Disease Free
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MabVax Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MV-0109DP001
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2016-12

CONDITIONS: Sarcoma
Keywords: Sarcoma; Metastatic; Vaccine; Adjuvant
MeSH Terms: conditions — Sarcoma; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Vaccine plus OPT-821
  Interventions: Biological: Trivalent ganglioside vaccine
- Arm B - OPT-821 immunologic adjuvant (Active Comparator): Patients will be given 10 injections of OPT-821 alone as a 1.0 ml subcutaneous injection in an outpatient setting at Visit Weeks 1, 2, 3, 8, 16, 28, 40, 52, 68 and 84
  Interventions: Biological: OPT-821

INTERVENTIONS:
Biological: Trivalent ganglioside vaccine — Patients will be given 10 injections of ganglioside vaccine plus adjuvant OPT-821 as a 1.0 ml subcutaneous injection in an outpatient setting at Visit Weeks 1, 2, 3, 8, 16, 28, 40, 52, 68 and 84
  Other Names: Trivalent ganglioside vaccine plus adjuvant OPT-821
  Arms: Arm A
Biological: OPT-821 — Patients will be given 10 injections of adjuvant OPT-821 as a 1.0 ml subcutaneous injection in an outpatient setting at Visit Weeks 1, 2, 3, 8, 16, 28, 40, 52, 68 and 84
  Other Names: Immunologic adjuvant OPT-821
  Arms: Arm B - OPT-821 immunologic adjuvant

SUMMARY:
Sarcoma patients are at high risk for their cancer to recur even when the sarcoma has been removed surgically or treated with radiation or chemotherapy. The patients in the study will be randomized (like flipping a coin) to receive either a vaccine that is combined with an immune system stimulant or the immune system stimulant alone. The immune system stimulant is called OPT-821 and is an immunological booster. The trivalent vaccine is being developed to teach the patient's immune system to recognize 3 types of sugars called GM2, GD2 and GD3 that are found primarily on the surface of sarcoma cells. If the trivalent vaccine can stimulate the patient's immune system to develop antibodies which recognize and target the GM2, GD2 and GM3 sugars, then the patient's antibodies could attack and kill any remaining sarcoma cells potentially preventing the recurrence of sarcoma.

DETAILED DESCRIPTION:
This study is a Phase II randomized, double-blind, multi-center study of a trivalent ganglioside vaccine plus the immunological adjuvant OPT-821 (Arm A) versus OPT-821 alone (Arm B) for patients with metastatic sarcoma at initial presentation or with relapsed disease who have been rendered disease-free following either surgical resection or multi-modality therapy. The primary aim of this study is to demonstrate the efficacy of vaccine therapy over non-specific immune therapy. Another aim of this study is to obtain sufficient data to further the development of this specific vaccine therapy as well as guide future study designs for therapeutic cancer vaccines in general.

To be eligible, patients must have histologically confirmed sarcoma, must be clinically free of disease after surgery or multimodality therapy, and must be within 8 weeks of completion of such therapy. Given the limited data regarding ganglioside expression in Ewing sarcoma, rhabdomyosarcoma, and gastrointestinal stromal tumors, patients with these sarcoma subtypes with the exception of pleomorphic/anaplastic rhabdomyosarcoma will be excluded. Patients must have a history of distant metastatic disease; patients with locally recurrent disease only will not be eligible, as these patients demonstrate a different natural history from those with metastatic disease.

All treatment will be performed in the outpatient setting. Patients will be randomized in a 1:1 ratio to receive a total of 10 treatments of either the vaccine plus OPT-821 (Arm A) or OPT-821 alone (Arm B). Treatment will be administered on Visit Weeks 1, 2, 3, 8, 16, 28, 40, 52, 68, and 84. All patients will receive 150 mcg of OPT-821.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 16 years or older.
2. American Joint Committee on Cancer (AJCC) Stage IV sarcoma with no current radiological evidence of residual disease following either surgery alone or multi-modality therapy for treatment of metastatic or relapsed disease. Patients must have presented with either newly diagnosed metastatic sarcoma or distant relapsed disease. Patients who present with more than one site of metastases are eligible as long as at least one new site is distant from the original site and the surgical resection(s) results in clear margins as assessed by the site pathologist. Non-surgical local ablative therapies such as SRS or cryotherapy cannot replace surgical resection of disease for the purpose of eligibility.
3. Histological confirmation of sarcoma, as performed by a pathologist at one of the participating study sites, prior to entry on study.
4. Patients must have undergone surgical metastectomy within 8 weeks prior to initiation of treatment on this study.
5. Patients previously treated with neoadjuvant chemotherapy and/or radiotherapy as part of a multi-modality treatment for metastatic disease must have recovered from all adverse effects of treatment and have returned to baseline status.
6. Imaging study performed within 4 weeks prior to administration of first vaccination documenting that patient has no evidence of disease. Study must include CT scan of chest, abdomen, and pelvis.
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1.
8. Weight ≥ 40 kg.
9. Have organ and marrow function as defined below:

   WBC ≥ 3.0 cells/mm3 Platelets ≥ 100,000/mm3 Total bilirubin ≤ 2.0 mg/dL AST (SGOT)/ALT (SGPT) ≤ 1.5 x ULN
10. Current use of an acceptable form of birth control.
11. Ability to understand English and to provide written informed consent and authorization for protected health information disclosure whether by self or by legally authorized representative.

Exclusion Criteria:

1. Patients with evidence of local or metastatic disease or who are not disease free at the time of the first vaccination.
2. Patients who develop locally recurrent disease only with no evidence of concurrent or previous distant metastatic disease. Patients with a primary retroperitoneal and/or uterine sarcoma that present with recurrence within the retroperitoneum or pelvis only are not eligible. Patients must have evidence of hematogenously disseminated distant disease.
3. Patients with brain or bone metastasis even if they are able to undergo complete surgical resection.
4. Patients with Ewing sarcoma, rhabdomyosarcoma (except for pleomorphic/anaplastic rhabdomyosarcoma), or gastrointestinal stromal tumors. Patients with pleomorphic/anaplastic rhabdomyosarcoma are eligible.
5. Patients previously treated with KLH or ganglioside containing vaccines or monoclonal antibodies (mAbs) against gangliosides.
6. Females of childbearing potential that are pregnant or intend to become pregnant or who are breastfeeding. Females must have negative βHCG test within two weeks of first vaccination.
7. Current active malignancy or history of malignancy, other than sarcoma, within the past two years, except for cervical carcinoma in situ or superficial skin cancer that has been surgically removed.
8. Any medical condition that may limit the ability of the patient to complete the full course of treatment or to respond immunologically to vaccination, (including autoimmune or neurodegenerative disorders such as multiple sclerosis and amyotrophic lateral sclerosis).
9. Patients requiring continuous doses of anti-inflammatory medications (steroids including inhaled steroids, non-steroidal anti-inflammatory drugs, or full dose aspirin). Episodic use of steroids or non-steroidal anti-inflammatory drugs permitted as long as they are not given within one week prior to or following vaccine administration. Continuous dosing of low-dose aspirin (≤ 81 mg/day) is acceptable.
10. Use of or treatment with a drug that has not received regulatory approval or participation in a drug or device study during the 28 days preceding the first vaccination.
11. Known history of HIV-positivity OR serologic evidence of HIV at screening or any immunodeficiency disorders or illnesses. Serologic positivity for the Hepatitis B Virus (HBV) or the Hepatitis C Virus (HCV), unless explained by a documented vaccination.
12. Inability or unwillingness to meet the attendance requirements of the study.
13. Any clinically significant abnormal finding at Screening (as determined by the principal investigator, in consultation with the Medical Monitor and the Sponsor), that would interfere with study participation, that would interfere with the evaluation or quality of the data, or that would put the patient at increased risk of illness or injury.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2010-06; Primary Completion 2013-09 (Actual); Study Completion 2017-03-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tap, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (13):
- United States (13):
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado (Denver), Denver, Colorado
  - Winship Cancer Institute at Emory Midtown, Atlanta, Georgia
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - University of Iowa Hospitals and Clinic, Iowa City, Iowa
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Hospital, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Oregon Health & Sciences University, Portland, Oregon
  - University of Pittsburg Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Fred Hutchinson Cancer Research Center/Seattle Cancer Care, Seattle, Washington

REFERENCES:
- [Derived] Rosenbaum E, Chugh R, Ryan CW, Agulnik M, Milhem MM, George S, Jones RL, Chmielowski B, Van Tine BA, Tawbi H, Elias AD, Read WL, Budd GT, Qin LX, Rodler ET, Hirman J, Weiden P, Bennett CM, Livingston PO, Ragupathi G, Hansen D, D'Angelo SP, Tap WD, Schwartz GK, Maki RG, Carvajal RD. A randomised phase II trial of a trivalent ganglioside vaccine targeting GM2, GD2 and GD3 combined with immunological adjuvant OPT-821 versus OPT-821 alone in metastatic sarcoma patients rendered disease-free by surgery. Eur J Cancer. 2022 Nov;176:155-163. doi: 10.1016/j.ejca.2022.09.003. Epub 2022 Oct 8. PMID 36215947
- [Derived] Cheung IY, Cheung NV, Modak S, Mauguen A, Feng Y, Basu E, Roberts SS, Ragupathi G, Kushner BH. Survival Impact of Anti-GD2 Antibody Response in a Phase II Ganglioside Vaccine Trial Among Patients With High-Risk Neuroblastoma With Prior Disease Progression. J Clin Oncol. 2021 Jan 20;39(3):215-226. doi: 10.1200/JCO.20.01892. Epub 2020 Dec 16. PMID 33326254
- See also: NCI sarcoma information — http://www.cancer.gov/cancertopics/types/soft-tissue-sarcoma
- See also: Related Info — http://www.mskcc.org/mskcc/html/435.cfm

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A- Vaccine Plus OPT-821: Trivalent ganglioside vaccine: Patients will be given 10 injections of ganglioside vaccine plus adjuvant OPT-821 as a 1.0 ml subcutaneous injection in an outpatient setting at Visit Weeks 1, 2, 3, 8, 16, 28, 40, 52, 68 and 84
Period: Overall Study
Arm/Group | Arm A- Vaccine Plus OPT-821 | Arm B - OPT-821 Immunologic Adjuvant
Started | 68 | 68
Completed | 20 | 21
Not Completed | 48 | 47

BASELINE CHARACTERISTICS:
Population: Adults (male or female), 16 years of age and older who have metastatic sarcoma at initial presentation or who had relapsed disease and are rendered disease-free following surgical metastectomy
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A- Vaccine Plus OPT-821 | Arm B - OPT-821 Immunologic Adjuvant | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 57 | 51 | 108
  >=65 years | 11 | 17 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 36 | 65
  Male | 39 | 32 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 62 | 61 | 123
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: The primary objective is to compare the progression-free survival (PFS) over time.
  Progression free survival is defined as the time from randomization until any evidence of tumor growth or appearance anywhere in the body or death from any cause as determined by the principal investigator at each site. The principal investigator will determine Progression-free survival by using CT scans to evaluate disease recurrence. For the purpose of this study, progression of disease is defined as the development of tumor growth or recurrence at any site of the body as determined by the principal investigator at each study site or death from disease
Time Frame: 3-years
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Arm A- Vaccine Plus OPT-821 | Arm B - OPT-821 Immunologic Adjuvant
Number analyzed (Participants) | 68 | 68
Days | 186 [163 to 193] | 271 [186 to 273]

2. Secondary Outcome: Overall Survival
Description: To compare the overall survival over time, to estimate the median and 3-year progression-free survival.
Time Frame: Measured over time
Reporting Status: Not Posted, anticipated posting 2017-04

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Arm A- Vaccine Plus OPT-821 | Arm B - OPT-821 Immunologic Adjuvant
Serious Adverse Events (participants affected / at risk) | 4/68 | 8/68
Other Adverse Events (participants affected / at risk) | 1/68 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Vaccine Plus OPT-821 (N=68) | Arm B - OPT-821 Immunologic Adjuvant (N=68)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — erythema left thigh. Possibly related, resolved.
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Not related, resolved.
Catheter site cellulitis (Infections and infestations) | 0 (0) | 1 (1) — Occurred 1 months after patient discontinued, unrelated and resolved.
Cerebrovascular Accident (Nervous system disorders) | 0 (0) | 1 (1) — Patient had numbness and weakness in the left upper extremity and a facial droop, symptoms resolved same day. Resolved, not related.
Anaphylactoid reaction (Immune system disorders) | 1 (1) | 0 (0) — chest and through tightness. Related, resolved
Hip Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) — Fracture of left hip. Not related, resolved.
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) — Not related, resolved
Cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1) — Not related, resolved
Death (General disorders) | 1 (1) | 0 (0) — Sudden death in patient with metastatic sarcoma and clinically unlikely to be related to the study drug.
Mitral valve disease (Cardiac disorders) | 0 (0) | 1 (1) — Not related, resolve.
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) — Possibly related. Resolved
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) — possibly related, resolved.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A- Vaccine Plus OPT-821 (N=68) | Arm B - OPT-821 Immunologic Adjuvant (N=68)
Ear infection (Infections and infestations) | 1 (1) | 0 (0) — Not Related, resolved

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site shall withhold publication of Site's individual Study results for a period of 18 months following completion of the Study at all sites, or until after Sponsor's written confirmation that Sponsor will not publish a joint, multicenter publication, whichever occurs first.